CLINICAL TRIAL: NCT00737893
Title: Erythropoietin to Enhance Recovery of Erectile Function in Men Following Radical Prostatectomy: a Prospective Randomized Controlled Trial (ERECT)
Brief Title: Erythropoietin to Enhance Recovery of Erectile Function in Men Following Radical Prostatectomy
Acronym: ERECT
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: IRB00048594; ERECT, EPO (Other: Johns Hopkins Brady Urological Institute)
Record Dates: First submitted 2008-08-19; First posted 2008-08-20 (Estimated); Results first posted 2020-08-13 (Actual); Last update posted 2021-04-08 (Actual); Status verified 2020-07

CONDITIONS: Prostate Cancer; Erectile Dysfunction
Keywords: Erythropoietin; Radical Prostatectomy; Erectile Dysfunction; Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms; Erectile Dysfunction | interventions — Erythropoietin

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Erythropoietin (EPO) (Experimental): 20,000 units of EPO given on the day before surgery, the day of surgery, and the day after surgery.
  Interventions: Drug: Erythropoietin (EPO)
- Placebo (Placebo Comparator): Placebo doses given the day before surgery, the day of surgery, and the day after surgery.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Placebo — Saline injection (solution prepared by research pharmacy) subcutaneously given the day before surgery, day of surgery, and the day after surgery.
  Arms: Placebo
Drug: Erythropoietin (EPO) — Erythropoietin (EPO)-induced Protein 29, Human; 20,000 units subcutaneously given the day before surgery, day of surgery, and the day after surgery.
  Arms: Erythropoietin (EPO)

SUMMARY:
This research study aims to explore the effectiveness of human erythropoietin versus placebo in promoting the recovery of erectile function in patients undergoing bilateral nerve-sparing radical retropubic prostatectomy for clinically localized prostate cancer.

Pre-clinical studies have shown erythropoietin potently promoted recovery of erectile function in rats and humans have similar receptors on penile tissues and the periprostatic neurovascular bundles. A clinical non-randomized study conducted in men undergoing radical prostatectomy demonstrated a benefit to recovery of erectile function.

Therefore, the hypothesis is that erythropoietin offers nerve protection in men undergoing nerve-sparing radical prostatectomy and results in a reduced degree of erectile dysfunction and also an improved rate of erection recovery following surgery.

DETAILED DESCRIPTION:
This study will evaluate the effectiveness of erythropoietin versus placebo in the recovery of erectile function in patients undergoing bilateral nerve-sparing radical prostatectomy for prostate cancer.

Recent laboratory findings in rat models and on human urogenital tissues suggest that erythropoietin may play a role in protection of the cavernous nerves during surgery. Some degree of nerve trauma occurs during bilateral nerve-sparing radical prostatectomy, but for most it is temporary. Erythropoietin will be studied as an investigational drug for enhancement of erectile function postoperatively in a prospective, randomized study. Erythropoietin has been used in many men undergoing open radical prostatectomy in the past according to FDA indications for preparation for noncardiac, nonvascular surgery with a high risk of blood loss. Evidence also suggests it is safe with no demonstration of increased risk of venous thromboembolism (blood clots) or cardiac events for men with prostate cancer undergoing radical prostatectomy.

The length of the study is 12 months and involves receiving a dose of study drug or placebo on the day before surgery, the day of surgery, and the day following surgery. The dose is given by subcutaneous injection. The study will also require the completion of questionnaires which will be completed online every three months until study completion (at 3, 6, 9, and 12 months) to assess outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Patient eligibility consists of men 40 to 65 years of age
* Localized prostate cancer

  * clinical stage T2a or lower
  * Gleason grade of 3+4 or 3+3
  * prostate specific antigen (PSA) < 10
* Scheduled to undergo curative prostatectomy applying bilateral nerve-sparing procedure, with intact pre-surgical erectile function
* International Index of Erectile Function-5 (IIEF-5) score of 22-25.
* The patient has a sexual partner, of at least 6 months.
* The patient's pre-surgical hematocrit is ≤ 48.
* The patient is willing to attempt intercourse at least 5 times per month following recovery from surgery.

Exclusion Criteria:

* The patient has known penile deformity or a history of Peyronie's disease.
* The patient has planned pre or post operative androgen therapy.
* The patient has planned pre or post operative radiation therapy.
* The patient is on anticoagulation therapy.
* The patient has a history of sickle cell anemia.
* The patient has a history of high or low blood pressure that is not controlled.
* The patient is taking medications called "nitrates"
* The patient has a history of heart problems such as angina, heart failure, irregular heartbeats, or myocardial infarction
* The patient has a history of history of drug or alcohol abuse.
* The patient currently smokes or has a 20 pack/year history of cigarette smoking.
* The patient has a history of acute or chronic depression
* The patient has a history liver problems, or kidney problems.
* The patient has a history of retinitis pigmentosa or severe vision loss, including a condition called NAION, Nonarteritic Anterior Ischemic Optic Neuropathy.
* The patient has a history of spinal trauma or surgery to the brain or spinal cord.
* The patient has contraindications to the use of phosphodiesterase type 5 (PDE 5) inhibitors.
* Patient is currently participating in another clinical investigation that would serve as a contraindication to administering erythropoietin.

Ages: 40 Years to 65 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 56 (Actual)
Dates: Start 2017-07-01 (Actual); Primary Completion 2019-12-31 (Actual); Study Completion 2019-12-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mohamad E Allaf, MD, Principal Investigator — Johns Hopkins Hospital - Brady Urological Institute
Locations (1):
- Johns Hopkins Hospital, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Patel HD, Allaf ME. Erythropoietin to Enhance Recovery of Erectile Function in Men Following Radical Prostatectomy: The ERECT Trial. Eur Urol Focus. 2019 Jul;5(4):698-699. doi: 10.1016/j.euf.2018.01.002. Epub 2018 Jan 17. PMID 29373284
- [Background] Allaf ME, Hoke A, Burnett AL. Erythropoietin promotes the recovery of erectile function following cavernous nerve injury. J Urol. 2005 Nov;174(5):2060-4. doi: 10.1097/01.ju.0000176808.94610.dd. PMID 16217394
- [Background] Liu T, Allaf ME, Lagoda G, Burnett AL. Erythropoietin receptor expression in the human urogenital tract: immunolocalization in the prostate, neurovascular bundle and penis. BJU Int. 2007 Nov;100(5):1103-6. doi: 10.1111/j.1464-410X.2007.07194.x. Epub 2007 Sep 14. PMID 17868418
- [Background] Burnett AL, Allaf ME, Bivalacqua TJ. Erythropoietin promotes erection recovery after nerve-sparing radical retropubic prostatectomy: a retrospective analysis. J Sex Med. 2008 Oct;5(10):2392-8. doi: 10.1111/j.1743-6109.2008.00980.x. Epub 2008 Sep 5. PMID 18778310
- [Result] Patel HD, Schwen ZR, Campbell JD, Gorin MA, Partin AW, Burnett AL, Allaf ME. Effect of Erythropoietin on Erectile Function after Radical Prostatectomy: The ERECT Randomized Clinical Trial. J Urol. 2021 Jun;205(6):1681-1688. doi: 10.1097/JU.0000000000001586. Epub 2021 Feb 3. PMID 33530745
- See also: The preoperative use of erythropoietin stimulating proteins prior to radical prostatectomy is not associated with increased cardiovascular or thromboembolic morbidity or mortality. — https://www.ncbi.nlm.nih.gov/pubmed/20513505
- See also: Preoperative recombinant human erythropoietin injection versus preoperative autologous blood donation in patients undergoing radical retropubic prostatectomy. — https://www.ncbi.nlm.nih.gov/pubmed/9372883

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Erythropoietin (EPO) | Placebo
Started | 29 | 27
Completed | 29 | 27
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Erythropoietin (EPO) | Placebo | Total
Number analyzed (Participants) | 29 | 27 | 56
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 54 [51 to 60] | 57 [52 to 61] | 55.5 [51.5 to 60]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 29 | 27 | 56
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 2 | 5 | 7
  White | 26 | 22 | 48
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 29 | 27 | 56

OUTCOME MEASURES:

1. Primary Outcome: Erectile Function as Assessed by the International Index of Erectile Function (IIEF) Questionnaire Erectile Function Domain
Description: Survey measuring erectile function using the IIEF (erectile function domain only) with overall score ranging from 0 to 30 where higher scores represent better erectile function.
Time Frame: At 6 months post-surgery
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Erythropoietin (EPO) | Placebo
Number analyzed (Participants) | 29 | 27
score on a scale | 14 [6.5 to 24] | 19 [8 to 23]

2. Secondary Outcome: Erectile Function as Assessed by the IIEF Questionnaire Erectile Function Domain
Description: as for outcome 1
Time Frame: At 3 months post-surgery
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Erythropoietin (EPO) | Placebo
Number analyzed (Participants) | 29 | 27
score on a scale | 11 [6 to 22] | 14 [6 to 23]

3. Secondary Outcome: Erectile Function as Assessed by the IIEF Questionnaire Erectile Function Domain
Description: as for outcome 1
Time Frame: At 9 months post-surgery
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Erythropoietin (EPO) | Placebo
Number analyzed (Participants) | 29 | 27
score on a scale | 20 [8 to 27] | 25 [12 to 28]

4. Secondary Outcome: Erectile Function as Assessed by the IIEF Questionnaire Erectile Function Domain
Description: as for outcome 1
Time Frame: At 12 months post-surgery
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Erythropoietin (EPO) | Placebo
Number analyzed (Participants) | 29 | 27
score on a scale | 22 [15.5 to 26] | 28 [18 to 30]

5. Secondary Outcome: Patient Score on the Overall IIEF Questionnaire
Description: Survey measuring erectile function using the IIEF (overall questionnaire) with overall score ranging from 0 to 75 where higher scores represent better erectile function.
Time Frame: At 3 months post-surgery
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Erythropoietin (EPO) | Placebo
Number analyzed (Participants) | 29 | 27
score on a scale | 33 [21 to 55] | 40 [21 to 53]

6. Secondary Outcome: Patient Score on the Overall IIEF Questionnaire
Description: as for outcome 5
Time Frame: At 6 months post-surgery
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Erythropoietin (EPO) | Placebo
Number analyzed (Participants) | 29 | 27
score on a scale | 37.5 [28.5 to 52] | 51 [32 to 55]

7. Secondary Outcome: Patient Score on the Overall IIEF Questionnaire
Description: as for outcome 5
Time Frame: At 9 months post-surgery
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Erythropoietin (EPO) | Placebo
Number analyzed (Participants) | 29 | 27
score on a scale | 50 [30 to 59] | 55 [33 to 66]

8. Secondary Outcome: Patient Score on the Overall IIEF Questionnaire
Description: as for outcome 5
Time Frame: At 12 months post-surgery
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Erythropoietin (EPO) | Placebo
Number analyzed (Participants) | 29 | 27
score on a scale | 53 [39 to 62] | 60.5 [44 to 68]

9. Secondary Outcome: Patient Score on Health-related Quality of Life Questionnaires (SF-12 MCS)
Description: Mental health composite score (MCS) component of the 12-Item Short Form Survey Instrument (SF-12) measured on a normalized scale with mean 50 and standard deviation 10 in the United States population. Higher scores represent a higher level of mental health.
Time Frame: At 3 months post-surgery
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Erythropoietin (EPO) | Placebo
Number analyzed (Participants) | 29 | 27
score on a scale | 54.9 [51.9 to 55.9] | 55.9 [44.8 to 57.7]

10. Secondary Outcome: Patient Score on Health-related Quality of Life Questionnaires (SF-12 MCS)
Description: as for outcome 9
Time Frame: At 6 months post-surgery
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Erythropoietin (EPO) | Placebo
Number analyzed (Participants) | 29 | 27
score on a scale | 55.9 [49.4 to 58.3] | 55.0 [50.6 to 57.8]

11. Secondary Outcome: Patient Score on Health-related Quality of Life Questionnaires (SF-12 MCS)
Description: as for outcome 9
Time Frame: At 9 months post-surgery
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Erythropoietin (EPO) | Placebo
Number analyzed (Participants) | 29 | 27
score on a scale | 55.9 [49.5 to 57.8] | 53.8 [51.1 to 57.8]

12. Secondary Outcome: Patient Score on Health-related Quality of Life Questionnaires (SF-12 MCS)
Description: as for outcome 9
Time Frame: At 12 months post-surgery
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Erythropoietin (EPO) | Placebo
Number analyzed (Participants) | 29 | 27
score on a scale | 55.3 [51.8 to 57.5] | 55.9 [51.4 to 57.9]

13. Secondary Outcome: Patient Score on the Expanded Prostate Cancer Index Composite (EPIC) Sexual Domain
Description: Sexual health domain score of the EPIC survey measuring health-related quality of life with higher scores representing better sexual function on a scale of 0 to 100.
Time Frame: At 3 months post-surgery
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Erythropoietin (EPO) | Placebo
Number analyzed (Participants) | 29 | 27
score on a scale | 43.6 [28.2 to 68.6] | 49.4 [31.4 to 63.5]

14. Secondary Outcome: Patient Score on the Expanded Prostate Cancer Index Composite (EPIC) Sexual Domain
Description: as for outcome 13
Time Frame: At 6 months post-surgery
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Erythropoietin (EPO) | Placebo
Number analyzed (Participants) | 29 | 27
score on a scale | 47.8 [35.9 to 65.1] | 53.2 [37.8 to 72.5]

15. Secondary Outcome: Patient Score on the Expanded Prostate Cancer Index Composite (EPIC) Sexual Domain
Description: as for outcome 13
Time Frame: At 9 months post-surgery
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Erythropoietin (EPO) | Placebo
Number analyzed (Participants) | 29 | 27
score on a scale | 59.6 [41.7 to 75] | 70.5 [37.8 to 80.8]

16. Secondary Outcome: Patient Score on the Expanded Prostate Cancer Index Composite (EPIC) Sexual Domain
Description: as for outcome 13
Time Frame: At 12 months post-surgery
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Erythropoietin (EPO) | Placebo
Number analyzed (Participants) | 29 | 27
score on a scale | 62.2 [46.5 to 77.9] | 73.7 [48.1 to 86.5]

17. Secondary Outcome: Patient Score on the Quality of Erection Questionnaire (QEQ)
Description: Survey measuring quality of erections using the QEQ with an overall score range of 0 to 100 where higher scores represent better erection quality.
Time Frame: At 3 months post-surgery
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Erythropoietin (EPO) | Placebo
Number analyzed (Participants) | 29 | 27
score on a scale | 20.8 [0 to 70.8] | 37.5 [0 to 70.8]

18. Secondary Outcome: Patient Score on the Quality of Erection Questionnaire (QEQ)
Description: as for outcome 17
Time Frame: At 6 months post-surgery
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Erythropoietin (EPO) | Placebo
Number analyzed (Participants) | 29 | 27
score on a scale | 37.5 [0 to 70.8] | 45.8 [0 to 75]

19. Secondary Outcome: Patient Score on the Quality of Erection Questionnaire (QEQ)
Description: as for outcome 17
Time Frame: At 9 months post-surgery
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Erythropoietin (EPO) | Placebo
Number analyzed (Participants) | 29 | 27
score on a scale | 66.7 [4.2 to 79.2] | 70.8 [20.8 to 87.5]

20. Secondary Outcome: Patient Score on the Quality of Erection Questionnaire (QEQ)
Description: as for outcome 17
Time Frame: At 12 months post-surgery
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Erythropoietin (EPO) | Placebo
Number analyzed (Participants) | 29 | 27
score on a scale | 70.8 [22.9 to 85.4] | 79.2 [41.7 to 100]

21. Secondary Outcome: Hemoglobin Level at 2 Weeks After Surgery
Description: Hemoglobin level at 2 weeks after surgery in grams per deciliter (g/dl).
Time Frame: 2 weeks after surgery
Measure: Median (Inter-Quartile Range); unit: g/dl
Arm/Group | Erythropoietin (EPO) | Placebo
Number analyzed (Participants) | 29 | 27
g/dl | 14.7 [14.1 to 15.2] | 13.6 [13.1 to 14.4]

22. Secondary Outcome: Number of Participants Requiring Transfusion During Hospitalization
Description: Assess the number of participants requiring transfusion during hospitalization.
Time Frame: During hospital stay, up to 1 week
Measure: Count of Participants; unit: Participants
Arm/Group | Erythropoietin (EPO) | Placebo
Number analyzed (Participants) | 29 | 27
Participants | 0 | 0

ADVERSE EVENTS:
Time Frame: 1 year
Description: Clavien-Dindo Complications (graded I, II, III, IV, and V) after surgery were assessed for all patients during hospitalization, at clinical follow-up visits, and via study survey follow-up. Clavien III or higher complications were considered serious.
Arm/Group | Erythropoietin (EPO) | Placebo
All-Cause Mortality (participants affected / at risk) | 0/29 | 0/27
Serious Adverse Events (participants affected / at risk) | 1/29 | 1/27
Other Adverse Events (participants affected / at risk) | 0/29 | 3/27
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Erythropoietin (EPO) (N=29) | Placebo (N=27)
Clavien III (Surgical and medical procedures) | 1 (1) | 1 (1) — Clavien III complication requiring procedure
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Erythropoietin (EPO) (N=29) | Placebo (N=27)
Clavien I-II (Surgical and medical procedures) | 0 (0) | 3 (3) — Clavien I-II complication

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-03-16): https://cdn.clinicaltrials.gov/large-docs/93/NCT00737893/Prot_SAP_000.pdf